CLINICAL TRIAL: NCT05502094
Title: Identification of the Effects of Post Covid Syndrome on the Autonomic Nervous System With Heart Rate Variability
Brief Title: Autonomic Nervous System Affection Due to Post Covid Syndrome
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Principle İnvestigator, Bahçeşehir University
Other Study IDs: STUDYAV0002
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Long Covid19; Autonomic Dysfunction
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Participants who experienced Post-Covid 19 syndrome were involved in this group.
  Interventions: Other: Heart Rate Variability Measurement
- Group 2: Participants who fully recovered after Covid-19 were involved in this group.
  Interventions: Other: Heart Rate Variability Measurement
- Group 3: Participants who had never had Covid-19 were involved in this group.
  Interventions: Other: Heart Rate Variability Measurement

INTERVENTIONS:
Other: Heart Rate Variability Measurement — The heart rate variability of the participants will be measured with the Polar H10 device with a measurement time of 5 minutes.

SUMMARY:
Post-Covid syndrome is defined as symptoms that develop in addition to respiratory symptoms in individuals who have had Covid-19 infection for more than 12 weeks. Symptoms such as fatigue, headache, cognitive impairment, dyspnea, heart palpitations, heat intolerance, digestive system disorders, sleep disorders, dermal problems, orthostatic intolerance come to the fore in individuals with post-Covid syndrome. It has been tried to be revealed in some studies that Covid-19 infection affects the autonomic nervous system (ANS) and the relationship between Post-Covid 19 syndrome and ANS dysfunction. Heart rate variability (HRV) measurement method can be used to evaluate ANS activity. HRV is a non-invasive method and is a measure of the change in heart rate over a period of time. HRV is a scalar quantity that shows the time between two beats of the heart and defines the oscillations between the R-R intervals. In HRV measurements, time-dependent and frequency-dependent measurement results are obtained and from these measurements, time-dependent RMSSD (square root of the square of the difference of the R-R intervals) and frequency-dependent high-frequency (HF) and low frequency (LF) measurement components are used in relation to the sympathetic nervous system (CNS) and parasympathetic nervous system (PSS). HRV can be measured in short-term (5 minutes) in terms of measurement time. The aim of this study is to clearly reveal the relationship between Post-Covid 19 syndrome and ANS dysfunction and to provide standardization related to HRV measurement method and sub-parameters.

DETAILED DESCRIPTION:
SARS-CoV-2 virus emerged with severe acute respiratory tract infection and pneumonia when turned into a chronic disease that can cause permanent symptoms in recovering individuals. Prolonged Covid-19 syndrome or Post-Covid 19 syndrome is defined as symptoms that develop in addition to respiratory symptoms in individuals who have had Covid-19 infection for more than 12 weeks. Symptoms such as fatigue, headache, cognitive impairment, dyspnea, heart palpitations, heat intolerance, digestive system disorders, sleep disorders, dermal problems, orthostatic intolerance come to the fore in individuals with post-Covid syndrome. It has been tried to be revealed in some studies that Covid-19 infection affects the autonomic nervous system (ANS) and the relationship between Post-Covid 19 syndrome and ANS dysfunction. It is known that the cytokine storm caused by Covid-19 is caused by sympathetic activation that induces the release of proinflammatory cytokines, and the virus is associated with autoantibodies such as α(alpha) and β(beta) adrenoceptors and muscarinic receptors and in this case it causes autoimmunological disorder and ANS dysfunction. ANS consists of craniosacral parasympathetic fibers and cervicothoracic sympathetic fibers and consists of a complex network structure that provides homeostasis of the body. The parasympathetic nervous system predominates in quiet "rest and digest" conditions, while the sympathetic nervous system drives the "fight or flight" response in stressful situations. Heart rate variability (HRV) measurement method can be used to evaluate ANS activity. HRV is a non-invasive method and is a measure of the change in heart rate over a period of time. HRV is a scalar quantity that shows the time between two beats of the heart and defines the oscillations between the R-R intervals. In HRV measurements, time-dependent and frequency-dependent measurement results are obtained and from these measurements, time-dependent RMSSD (square root of the square of the difference of the R-R intervals) and pNN50 (the proportionality coefficient obtained by dividing the total number of R-R intervals by NN50), frequency-dependent high-frequency (HF) and low frequency (LF) measurement components are used in relation to the sympathetic nervous system (CNS) and parasympathetic nervous system (PSS). HRV can be measured in 3 different ways, as ultra short-term (<5 minutes), short-term (5 minutes) and long-term (24 hours), in terms of measurement time, and these values provide different results from each other. While 24-hour long-term measurements are preferred in cardiac diseases with a risk of mortality, short-term and ultra short-term measurements may be preferred in measuring the effect of chronic and metabolic diseases on HRV. The aim of this study is to clearly reveal the relationship between Post-Covid 19 syndrome and ANS dysfunction and to provide standardization related to HRV measurement method and sub-parameters.

Our study in which investigated the effect of post-Covid 19 syndrome on the autonomic nervous system, will be carried out in the Bahçeşehir University Institute of Health Sciences. Written consent will be obtained from the participants, indicating that they agreed to participate in the study and the content of the study was presented verbally and in writing form. Patients will be taken a short 5-minute measurement for HRV measurement once during the study. Before the evaluation, sociodemographic information will be obtained from the participants in the form of a questionnaire and the symptoms experienced by the participants were recorded. Participants will be warned not to exert excessive effort and not to take any medication or treatment before the measurement. In the research form given to the patients, the symptoms of individuals with Post-Covid 19 syndrome will be marked and the percentage of these symptoms was calculated. These symptoms will be determined as fatigue, headache, cognitive impairment, dyspnea, heart palpitation, heat intolerance, digestive system disorders, sleep disturbance, dermal problems, orthostatic intolerance.

A total of 60 participants whom between the ages of 18-45 will include in our study, including 20 participants (n=20) who experience Post-Covid 19 syndrome, participants who fully recover after Covid-19 (n=20) and participants who has never have Covid-19 (n=20). In order for the study groups to be homogeneous, the ratio of the number of men and women in the groups will tried to be equal.

The Polar H10 wearable HRV measurement technology, which we use in our study and produced by Polar Electro company, is a device that helps to measure the R-R interval at rest and at different activity intensities (Picture 1). In the study conducted by Schweizer et al., it shows that the Polar H10 device had 99.6% R-R interval signal quality during 5 different activities (16).

In our research, the measurements will made with the Polar H10 device were analyzed on the computer with the Kubios Software 3.5.0 program (https://www.kubios.com). With this program, it is possible to apply time dependent, frequency dependent and nonlinear analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Participants who aged 18-45 years

Exclusion Criteria:

* Considering that the estrogen level in the body affects ANS among female patients, female participants in pre-menopausal, post-menopausal and pregnancy conditions
* Being in the date of women in the menstruation period
* Cancer diagnosis and treatment,
* Neurological disease diagnosis,
* Immunological disease diagnosis,
* History of cardiovascular disease diagnosis
* Presence of acute infection
* Participants who used medication in the last 6 months for the treatment of ANS dysfunction were also excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It consists of participants who have not had Covid 19 and who have and did not show prolonged symptoms afterward.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability-Time Dependent(RMSSD) | Through study completion, an average of 1 year.
  RMSSD: Root mean square of successive RR interval differences. Unit: miliseconds(ms)
Heart Rate Variability-Frequency Dependent- Low Frequency (LF) Power | Through study completion, an average of 1 year.
  Low Frequency Power (LF): Relative power of the low-frequency band (0.04-0.15 Hz) in normal units. Unit: nu
Heart Rate Variability-Frequency Dependent- High Frequency (HF) Power | Through study completion, an average of 1 year.
  High Frequency (HF) Power: Relative power of the high-frequency band (0.15-0.4 Hz) in normal units. Unit:nu
Heart Rate Variability-Frequency Dependent- High Frequency (HF)/ Low Frequency(HF/LF) | Through study completion, an average of 1 year.
  High Frequency (HF)/ Low Frequency(HF/LF): Ratio of LF-to-HF power. Unit: %

SECONDARY OUTCOMES:
Body mass index (BMI) | Through study completion, an average of 1 year.
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Veysel Özden, M.D., Study Director — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198
- [Result] National Insitute for Health and Care Excellence; SIGN. Royal College of General Practitioners COVID-19 Guideline Scope: Management of the Long-Term Effects of COVID-19; NICE: London, UK, 2020; pp. 1-7.
- [Result] Cares-Marambio K, Montenegro-Jimenez Y, Torres-Castro R, Vera-Uribe R, Torralba Y, Alsina-Restoy X, Vasconcello-Castillo L, Vilaro J. Prevalence of potential respiratory symptoms in survivors of hospital admission after coronavirus disease 2019 (COVID-19): A systematic review and meta-analysis. Chron Respir Dis. 2021 Jan-Dec;18:14799731211002240. doi: 10.1177/14799731211002240. PMID 33729021
- [Result] Konig MF, Powell M, Staedtke V, Bai RY, Thomas DL, Fischer N, Huq S, Khalafallah AM, Koenecke A, Xiong R, Mensh B, Papadopoulos N, Kinzler KW, Vogelstein B, Vogelstein JT, Athey S, Zhou S, Bettegowda C. Preventing cytokine storm syndrome in COVID-19 using alpha-1 adrenergic receptor antagonists. J Clin Invest. 2020 Jul 1;130(7):3345-3347. doi: 10.1172/JCI139642. No abstract available. PMID 32352407
- [Result] Goldstein DS. The extended autonomic system, dyshomeostasis, and COVID-19. Clin Auton Res. 2020 Aug;30(4):299-315. doi: 10.1007/s10286-020-00714-0. Epub 2020 Jul 22. PMID 32700055
- [Result] Dani M, Dirksen A, Taraborrelli P, Torocastro M, Panagopoulos D, Sutton R, Lim PB. Autonomic dysfunction in 'long COVID': rationale, physiology and management strategies. Clin Med (Lond). 2021 Jan;21(1):e63-e67. doi: 10.7861/clinmed.2020-0896. Epub 2020 Nov 26. PMID 33243837
- [Result] McCorry LK. Physiology of the autonomic nervous system. Am J Pharm Educ. 2007 Aug 15;71(4):78. doi: 10.5688/aj710478. PMID 17786266
- [Result] Tindle J, Tadi P. Neuroanatomy, Parasympathetic Nervous System. 2022 Oct 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK553141/ PMID 31985934
- [Result] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Result] Barauskiene V, Rumbinaite E, Karuzas A, Martinkute E, Puodziukynas A. Importance of Heart Rate Variability in Patients with Atrial Fibrillation. J Cardiol Clin Res. 2016;4:1080.
- [Result] Costa JYB, Anunciaçao PG, Ruiz RJ, Casonatto J, Polito MD. Effect of Caffeine Intake on Blood Pressure and Heart Rate Variability after a Single Bout of Aerobic Exercise. International SportMed Journal 2012; 13 (3): 109-121.
- [Result] Hayano J, Yuda E. Pitfalls of assessment of autonomic function by heart rate variability. J Physiol Anthropol. 2019 Mar 13;38(1):3. doi: 10.1186/s40101-019-0193-2. PMID 30867063
- [Result] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Result] Kleiger RE, Miller JP, Bigger JT Jr, Moss AJ. Decreased heart rate variability and its association with increased mortality after acute myocardial infarction. Am J Cardiol. 1987 Feb 1;59(4):256-62. doi: 10.1016/0002-9149(87)90795-8. PMID 3812275
- [Result] Gilgen-Ammann R, Schweizer T, Wyss T. RR interval signal quality of a heart rate monitor and an ECG Holter at rest and during exercise. Eur J Appl Physiol. 2019 Jul;119(7):1525-1532. doi: 10.1007/s00421-019-04142-5. Epub 2019 Apr 19. PMID 31004219